CLINICAL TRIAL: NCT00779090
Title: The Influence of a Functional Residual Capacity Guided Alveolar Recruitment Strategy After Open Endotracheal Suctioning on Oxygenation and Regional Ventilation
Brief Title: Functional Residual Capacity (FRC) Guided Alveolar Recruitment Strategy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Hermann Heinze, Department of Anaesthesiology, University of Lübeck, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FRCGARS-1
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Ventilation; Functional Residual Capacity
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A_RM (Experimental): Patients with FRC after open endotracheal suctioning of more than 94% of baseline randomized to receive an alveolar recruitment manoeuvre.
  Interventions: Procedure: Alveolar recruitment manoeuvre
- Group A_NRM (No Intervention): Patients with FRC after open endotracheal suctioning of more than 94% of baseline randomized to receive no alveolar recruitment manoeuvre.
- Group B_RM (Experimental): Patients with FRC after open endotracheal suctioning of less than 94% of baseline randomized to receive an alveolar recruitment manoeuvre.
  Interventions: Procedure: Alveolar recruitment manoeuvre
- Group B_NRM (No Intervention): Patients with FRC after open endotracheal suctioning of less than 94% of baseline randomized to receive no alveolar recruitment manoeuvre.

INTERVENTIONS:
Procedure: Alveolar recruitment manoeuvre — Increase airway pressure during pressure controlled ventilation up to peak-airway pressure of 40 cmH20 and PEEP of 15 cmH20.
  Arms: Group A_RM; Group B_RM

SUMMARY:
In ventilated patients open endotracheal suctioning may lead to alveolar derecruitment, which can be monitored by means of functional residual capacity (FRC) measurements. The investigators hypothesized that a recruitment strategy based on FRC measurements would improve oxygenation and regional ventilation after an open endotracheal suctioning manoeuvre.

DETAILED DESCRIPTION:
In mechanically ventilated patients the functional residual capacity will be measured before (baseline) and after an open endotracheal suctioning manoeuvre. Based on these changes patients will be divided into two groups: Group A with more than 94% of baseline FRC, and Group B with less than 94% of baseline FRC. Both groups will be randomized to receive an alveolar recruitment manoeuvre or no alveolar recruitment manoeuvre, leading to four groups. Oxygenation and regional ventilation with electrical impedance tomography will be studied.

ELIGIBILITY:
Inclusion Criteria:

* ventilated after elective cardiac surgery

Exclusion Criteria:

* hemodynamic instability (eg. intraaortic balloon pump)
* acute lung injury, i.e. PEEP > 10cmH20 or FiO2 > 0.4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Arterial oxygenation | 60 minutes

SECONDARY OUTCOMES:
Regional ventilation | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Heinze, MD, Principal Investigator — Department of Anaesthesiology, University of Lübeck

REFERENCES:
- [Derived] Heinze H, Eichler W, Karsten J, Sedemund-Adib B, Heringlake M, Meier T. Functional residual capacity-guided alveolar recruitment strategy after endotracheal suctioning in cardiac surgery patients. Crit Care Med. 2011 May;39(5):1042-9. doi: 10.1097/CCM.0b013e31820eb736. PMID 21336125